CLINICAL TRIAL: NCT00231114
Title: Safety and Effectiveness of the Alair® System for the Treatment of Asthma: A Multicenter Randomized Clinical Trial(Asthma Intervention Research (AIR2) Trial)
Brief Title: Asthma Intervention Research 2 (AIR2) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-02
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2010-11-29 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2014-03

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alair (Experimental): Treatment of airways with the Alair System
  Interventions: Device: Alair System
- Sham (Sham Comparator): Sham treatment of airways
  Interventions: Device: Alair System

INTERVENTIONS:
Device: Alair System — Treatment of airways with the Alair System
  Arms: Alair
Device: Alair System — Sham treatment of airways with the Alair System
  Arms: Sham

SUMMARY:
The objective of this randomized, double blind, sham-controlled study is to demonstrate the safety and effectiveness of the Alair System in a population of subjects with severe asthma who are still symptomatic despite being managed on conventional therapy of high doses of inhaled corticosteroids and long-acting β2-agonists.

The primary efficacy endpoint will be the difference between Study groups in the change in Asthma Quality of Life Questionnaire (AQLQ) score from Baseline and the average score from the 6-, 9-, and 12-month follow-up visits.

All other outcome measures assessed at 12 months post-treatment.

This will be a multicenter, randomized, double-blind, sham-controlled study comparing the effects of treatment with the Alair System to conventional therapy of inhaled corticosteroids (ICS) and long-acting β2-agonists (LABA).

A Bayesian adaptive approach to sample size selection is used with a randomization scheme of 2:1 (two Alair Group Subjects for every one Control Group Subject).

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult between the ages of 18 to 65 years.
* Subject has asthma and is taking regular maintenance medication that includes Inhaled corticosteroid (ICS) AND long acting ß2-agonist (LABA).
* Subject has a Pre-bronchodilator Forced Expiratory Volume in one second (FEV1) of greater than or equal to 60% of predicted after medication stabilization during the Baseline Period.
* Subject has a PC20 < 8 mg/ml per methacholine inhalation test using standardized methods. PC20 is a provocative concentration of Provocholine® (a brand of methacholine chloride) resulting in a drop of FEV1 of 20% or more from Baseline.
* Subject has at least two days of asthma symptoms during the 4-weeks of the Baseline Diary Period.
* Subject is a non-smoker for 1 year or greater (if former smoker, less than 10 pack years total smoking history).

Exclusion Criteria:

* Subject has a Post-bronchodilator FEV1 of less than 65%.
* Subject has 3 or more hospitalizations for exacerbations of asthma in the previous year; OR a history of life-threatening asthma, defined by past intubations for asthma, or ICU admission for asthma within the prior 24 months.
* Subject has a history of recurrent lower respiratory tract infections requiring antibiotics (more than 3 in the past 12 months).
* Subject has a history of recurrent oral steroid use for asthma (4 or more pulses of oral steroids in the past 12 months).
* Subject has a known sensitivity to medications required to perform bronchoscopy (such as lidocaine, atropine and benzodiazepines).
* Subject has known systemic hypersensitivity or contraindication to Methacholine chloride or other parasympathomimetic agents.
* Subject has other medical criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder S Shargill, PhD, Study Director — Asthmatx, Inc.
Locations (39):
- United States (22):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - University of Southern California, Adult Asthma and Allergy Center, Los Angeles, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Peoria Pulmonary Associates, Ltd., Peoria, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veritas Clinical Specialties, Topeka, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Womens's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - HealthPartners Specialty Center, Lung and Sleep Health, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Vincent Catholic Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennyslvania, Philadelphia, Pennsylvania
  - Clinical Research Solutions, PC - Baptist Hospitals of East Tennesse, Knoxville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Virginia Hospital Center, Arlington, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
- Australia (3):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
- Brazil (4):
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Irmandade Santa Casa de Miscericordia de Porto Alegre, Porto Alegre
  - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
  - Faculdade da Medicina do ABC, São Paulo
- Canada (3):
  - Firestone Institute of Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario
  - Montreal Chest Institute, McGill University, Montreal, Quebec
  - Hopital Laval, Centre de Pneumologie, Sainte-Foy, Quebec
- Odense Universitets Hospital, University of Odense, Odense, Denmark
- Universitair Medisch Centrum, Groningen, Netherlands
- United Kingdom (5):
  - Gartnavel General Hospital, University of Glasgow, Glasgow, Scotland
  - Birmingham Heartlands Hospital, Birmingham
  - Glenfield General Hospital, Univ. Hospitals of Leicester, Leicester
  - Chelsea & Westminster Healthcare NHS Trust, London
  - Northwest Lung Research Center, Univ. of Manchester, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pavord ID, Thomson NC, Niven RM, Corris PA, Chung KF, Cox G, Armstrong B, Shargill NS, Laviolette M; Research in Severe Asthma Trial Study Group. Safety of bronchial thermoplasty in patients with severe refractory asthma. Ann Allergy Asthma Immunol. 2013 Nov;111(5):402-7. doi: 10.1016/j.anai.2013.05.002. Epub 2013 Jun 13. PMID 24125149
- [Result] Wechsler ME, Laviolette M, Rubin AS, Fiterman J, Lapa e Silva JR, Shah PL, Fiss E, Olivenstein R, Thomson NC, Niven RM, Pavord ID, Simoff M, Hales JB, McEvoy C, Slebos DJ, Holmes M, Phillips MJ, Erzurum SC, Hanania NA, Sumino K, Kraft M, Cox G, Sterman DH, Hogarth K, Kline JN, Mansur AH, Louie BE, Leeds WM, Barbers RG, Austin JH, Shargill NS, Quiring J, Armstrong B, Castro M; Asthma Intervention Research 2 Trial Study Group. Bronchial thermoplasty: Long-term safety and effectiveness in patients with severe persistent asthma. J Allergy Clin Immunol. 2013 Dec;132(6):1295-302. doi: 10.1016/j.jaci.2013.08.009. Epub 2013 Aug 30. PMID 23998657
- [Result] Castro M, Rubin AS, Laviolette M, Fiterman J, De Andrade Lima M, Shah PL, Fiss E, Olivenstein R, Thomson NC, Niven RM, Pavord ID, Simoff M, Duhamel DR, McEvoy C, Barbers R, Ten Hacken NH, Wechsler ME, Holmes M, Phillips MJ, Erzurum S, Lunn W, Israel E, Jarjour N, Kraft M, Shargill NS, Quiring J, Berry SM, Cox G; AIR2 Trial Study Group. Effectiveness and safety of bronchial thermoplasty in the treatment of severe asthma: a multicenter, randomized, double-blind, sham-controlled clinical trial. Am J Respir Crit Care Med. 2010 Jan 15;181(2):116-24. doi: 10.1164/rccm.200903-0354OC. Epub 2009 Oct 8. PMID 19815809
- [Derived] Castro M, Rubin A, Laviolette M, Hanania NA, Armstrong B, Cox G; AIR2 Trial Study Group. Persistence of effectiveness of bronchial thermoplasty in patients with severe asthma. Ann Allergy Asthma Immunol. 2011 Jul;107(1):65-70. doi: 10.1016/j.anai.2011.03.005. Epub 2011 Apr 14. PMID 21704887
- See also: The AIR2 Extension Study (PAS1) contains the Year 2 to Year 5 Study Results. — http://clinicaltrials.gov/ct2/show/NCT01350414?term=PAS1&rank=1

RESULTS

PARTICIPANT FLOW:
Groups:
- Alair: Alair treatment plus conventional therapy with inhaled corticosteroids and long acting β2-agonists.
- Sham: Sham bronchoscopy plus conventional therapy with inhaled corticosteroids and long acting β2-agonists.
Period: Randomized
Arm/Group | Alair | Sham
Started | 196 | 101
Completed | 190 | 98
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 6 | 3
Period: Treatment Period
Arm/Group | Alair | Sham
Started | 190 | 98
Completed | 189 | 98
Not Completed | 1 | 0
Not completed — Death: Motor Vehicle Accident | 1 | 0
Period: Post-Treatment Period
Arm/Group | Alair | Sham
Started | 189 | 98
Completed | 181 | 97
Not Completed | 8 | 1
Not completed — Lost to Follow-up | 6 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alair | Sham | Total
Number analyzed (Participants) | 190 | 98 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.89) | 40.6 (11.85) | 40.65 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 60 | 169
  Male | 81 | 38 | 119
Region of Enrollment [Number; unit: participants]
  United States | 59 | 29 | 88
  Canada | 36 | 17 | 53
  Brazil | 55 | 29 | 84
  United Kingdom | 28 | 15 | 43
  Netherlands | 5 | 2 | 7
  Australia | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Integrated Asthma Quality of Life Questionnaire (AQLQ) Score (Change From Baseline)
Description: Change between Baseline and the average of 6-, 9-, and 12-month Follow-Up Visits. The AQLQ consists of 32 questions (scale from 1 to 7, where 7 reflects a higher quality of life). An increase in the AQLQ score indicates a better quality of life. The average of the 6-, 9-, and 12-month differences in the AQLQ Score are referred to as the "Integrated AQLQ Score."
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Units on a scale | 1.35 (1.10) | 1.16 (1.23)

2. Secondary Outcome: Percent Symptom-Free Days (Change From Baseline)
Description: Change between Baseline and 12-month Follow-Up Visit. Symptom-Free Days were defined as days when Subject reported no cough, wheeze, breathlessness, or sputum during the daytime, and no wheeze, cough, or awakenings due to asthma symptoms during nighttime.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Percent Change | 24.4 (36.16) | 21.0 (35.48)

3. Secondary Outcome: Total Symptom Score (Change From Baseline)
Description: Change from Baseline and 12-month Follow-Up Visit. Total Symptom Score comprises the sum of these six asthma symptom measurements: wheeze during the night, cough during the night, wheeze during the day, cough during the day, breathlessness during the day, and sputum production during the day. Each of these symptoms is scored on a scale of 0 to 3 each day by the subject. The sum of the scores for these 6 symptoms comprises the Total Symptom Score, which measures overall asthma symptoms. The maximum score possible is 18. A lower Total Symptom score represents better asthma control.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Units on a scale | -1.7 (2.32) | -1.6 (2.64)

4. Secondary Outcome: Number of Puffs of Rescue Medication Used (Change From Baseline)
Description: Change between Baseline and 12-Month Follow-up Visit. Average number of puffs per week. Rescue medications for asthma are short-acting beta-agonists that bring quick relief of asthma symptoms.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Puffs/7 Days
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Puffs/7 Days | -6.0 (16.67) | -4.3 (12.19)

5. Secondary Outcome: Percent Days Rescue Medication Used (Change From Baseline)
Description: Change between Baseline and 12-Month Follow-up Visit. Rescue medications for asthma are short-acting beta-agonists that bring quick relief of asthma symptoms.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Percent Change | -24.0 (33.51) | -22.0 (36.14)

6. Secondary Outcome: Asthma Control Questionnaire (ACQ) Score (Change From Baseline)
Description: Change between Baseline and 12-month Follow-Up Visit. The ACQ is a self-administered patient questionnaire that also includes the patient's FEV1 value (% Predicted) that assesses individual subject asthma control. The ACQ comprises 6 questions that relate to the patient's asthma symptoms, activity limitations, and daily rescue bronchodilator use, and FEV1. Each question is scored from 0 (Better) to 6 (Worse). A decrease in the ACQ score indicates better asthma control.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Units on a scale | -0.82 (0.95) | -0.77 (1.08)

7. Secondary Outcome: Morning Peak Expiratory Flow (amPEF) (Change From Baseline)
Description: Change between Baseline and 12-month Follow-Up Visit. The peak expiratory flow rate measures the maximal rate at which a person can exhale air.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: L/Min
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
L/Min | 27.8 (49.78) | 22.3 (51.54)

8. Secondary Outcome: Pre-Bronchodilator FEV1 (Percent Predicted) (Change From Baseline)
Description: Change between Baseline and 12-month Follow-Up Visit. The FEV1 is the volume of air expired during the first second of a maximal effort expiration started at total lung capacity.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Percent Change | -1.4 (14.71) | -0.1 (13.80)

9. Secondary Outcome: Post-Bronchodilator FEV1 (Percent Predicted) (Change From Baseline)
Description: as for outcome 8
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Percent Change | -2.8 (10.74) | -2.4 (8.33)

10. Other Pre Specified Outcome: Rate of Severe Exacerbations Requiring Systemic Corticosteroids
Description: Rate of occurrence of worsening of asthma requiring treatment with oral or intravenous corticosteroids, OR a doubling of the baseline inhaled corticosteroid dose for at least 3 days, OR any temporary increase in the dosage of oral corticosteroids for a Subject taking maintenance oral corticosteroids at Study entry.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Events/Subject/Year
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Events/Subject/Year | 0.48 (0.07) | 0.70 (0.12)

11. Other Pre Specified Outcome: Percentage of Subjects With Severe Exacerbations Requiring Systemic Corticosteroids
Description: Percent of subjects experiencing worsening of asthma requiring treatment with oral or intravenous corticosteroids, OR a doubling of the baseline inhaled corticosteroid dose for at least 3 days, OR any temporary increase in the dosage of oral corticosteroids for a Subject taking maintenance oral corticosteroids at Study entry.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Number; unit: Percent of Subjects
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Percent of Subjects | 26.3 | 39.8

12. Other Pre Specified Outcome: Days Lost From Work/School/Other Activities Due to Asthma
Time Frame: 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Days/Subject/Year
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Days/Subject/Year | 1.32 (0.36) | 3.9 (1.6)

13. Other Pre Specified Outcome: Unscheduled Physician Office Visits for Respiratory Symptoms
Time Frame: 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Events/Subject/Year
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Events/Subject/Year | 0.28 (0.05) | 0.36 (0.09)

14. Other Pre Specified Outcome: Emergency Room Visits for Respiratory Symptoms
Time Frame: 12 Months
Population: Intent-to-Treat (ITT) population. Consists of all randomized subjects who were administered at least one bronchoscopy.
Measure: Mean (Standard Deviation); unit: Events/Subject/Year
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Events/Subject/Year | 0.07 (0.03) | 0.43 (0.20)

15. Other Pre Specified Outcome: Hospitalizations for Respiratory Symptoms
Time Frame: 12 Months
Measure: Number; unit: Events/Subject/Year
Arm/Group | Alair | Sham
Number analyzed (Participants) | 190 | 98
Events/Subject/Year | 0.04 | 0.13

ADVERSE EVENTS:
Description: Rates in "Other Adverse Events" include Serious Adverse Events. Two subjects in the BT group did not complete the 6-week visit and were classified as having missed visits. These subjects were later classified as lost to follow-up or withdrawn. Conservatively, the lowest denominator (187 instead of 189) to estimate post-treatment risk has been used.
Groups:
- Alair (Treatment Period): Day of first bronchoscopy session until 6 weeks after the last bronchoscopy session. Airways treated with the Alair System.
- Sham (Treatment Period): Day of first bronchoscopy session until 6 weeks after the last bronchoscopy session. Sham treatment.
- Alair (Post-Treatment Period): Six weeks after the last bronchoscopy session until 12 Months. Airways treated with the Alair System.
- Sham (Post-Treatment Period): Six weeks after the last bronchoscopy session until 12 Months. Sham treatment.
Arm/Group | Alair (Treatment Period) | Sham (Treatment Period) | Alair (Post-Treatment Period) | Sham (Post-Treatment Period)
Serious Adverse Events (participants affected / at risk) | 19/190 | 4/98 | 12/187 | 10/98
Other Adverse Events (participants affected / at risk) | 176/190 | 82/98 | 157/187 | 86/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alair (Treatment Period) (N=190) | Sham (Treatment Period) (N=98) | Alair (Post-Treatment Period) (N=187) | Sham (Post-Treatment Period) (N=98)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthma (Multiple Symptoms) (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 5 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Forced Expiratory Volume Decreased (Investigations) | 1 | 0 | 0 | 0
Foreign Body Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haematoma Evacuation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alair (Treatment Period) (N=190) | Sham (Treatment Period) (N=98) | Alair (Post-Treatment Period) (N=187) | Sham (Post-Treatment Period) (N=98)
Acute Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7 | 8
Asthma (Multiple Symptoms) (Respiratory, thoracic and mediastinal disorders) | 99 | 38 | 51 | 42
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 6 | 6 | 5
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 13 | 5
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 17 | 10 | 3 | 1
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 26 | 13 | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 14 | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 6 | 4 | 1
Headache (Nervous system disorders) | 27 | 9 | 9 | 3
Influenza (Infections and infestations) | 8 | 2 | 8 | 12
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 15 | 2 | 6 | 6
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 20 | 5
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 1 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 5 | 4
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 8 | 6
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 12 | 7
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 2 | 3
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 38 | 11 | 56 | 25
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 11 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 29 | 6 | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less